CLINICAL TRIAL: NCT03210324
Title: Mifepristone Tablets in the Treatment of Symptomatic Uterine Fibroids With Safety and Efficacy in Open, Multicenter Phase IV Clinical Studies
Brief Title: A Study on the Mifepristone Tablets in the Treatment of Symptomatic Uterine Fibroids With Safety and Efficacy
Status: Terminated | Phase: Phase 4 | Type: Interventional
Why Stopped: It is difficult to recruit enough participants
Sponsor: China Resources Zizhu Pharmaceutical Co., Ltd. (Industry)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: ZZYY-MF-10-401
Record Dates: First submitted 2017-06-12; First posted 2017-07-06 (Actual); Last update posted 2019-08-07 (Actual); Status verified 2019-08

CONDITIONS: Uterine Fibroid
Keywords: mifepristone antiprogestins
MeSH Terms: conditions — Leiomyoma | interventions — Mifepristone

STUDY DESIGN:
Masking Description: Open Label
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- Mifepristone A group (Experimental): Mifepristone tablets for 12 weeks with two follow-up
  Interventions: Drug: Mifepristone tablets
- Mifepristone B group (Experimental): Mifepristone tablets for 12 weeks with four follow-up
  Interventions: Drug: Mifepristone tablets
- Mifepristone C group (Experimental): Mifepristone tablets for 24 weeks with four follow-up
  Interventions: Drug: Mifepristone tablets

INTERVENTIONS:
Drug: Mifepristone tablets — Daily 10mg, Po, Qd, each 10mg/tablets。Start from 1 to 3 days of the menstruation, take 1 tablet after 2 hours of fasting, and no eating for 2 hours after taking the pill. Group A and group B: treatment for 12 weeks, Group C: treatment for 24 weeks.

SUMMARY:
To investigate the efficacy and adverse effects of mifepristone tablets in widely used conditions, to evaluate the relationship between interests and risks used in general or special populations, to further observe the safety and efficacy of drugs.

DETAILED DESCRIPTION:
Uterine fibroids (also referred to as myomas, leiomyomas, leiomyomata, and fibromyomas) are non-cancerous (benign) tumors that grow within the muscle tissue of the uterus. Approximately 20-40% of women 35 years and older have fibroids. While many women with fibroids do not experience any symptoms, the location and size of fibroids can cause symptoms that can affect a woman's quality of life.

Fibroids are hormonally sensitive so symptoms are likely to be cyclical with menstruation. Fibroid growth is dependent on hormone levels; an increase in a woman's hormone levels may cause the size of fibroids to increase. During menopause, these hormones decrease dramatically and may cause fibroid symptoms to diminish.

Mifepristone is an antiestrogen hormone that antagonizes progesterone at receptor levels. Estrogen is generally considered to be a major contributor to uterine fibroids, but many studies have confirmed that progesterone can promote fibroid cell mitosis, and thus promote fibroids growth. In recent years, domestic and international clinical studies have shown that mifepristone treatment for 3 months can significantly reduce the size of uterine fibroids to achieve complete amenorrhea, improve bleeding caused by anemia, reduce clinical symptoms, uterine fibroids to reduce the size of complex Of the hysterectomy surgery into a simple, to avoid surgery caused by other organs of the injury, shorten the operation time, reduce the amount of surgical bleeding and blood transfusion, so that patients recover faster after surgery The literature reported the clinical use of 50mg, 25mg, 10mg and 5mg. The minimum dose of 10mg daily, 3 months can reduce the average size of uterine fibroids nearly half. Daily 5mg on fibroids shrink is not obvious. Mifepristone tablets is developed by the China Resources Zizhu Pharmaceutical Co., Ltd. Drugs and Drugs 1.6, each tablet 10mg, for adult age women have moderate to severe symptoms of uterine fibroids before the treatment of national food and drug supervision and management General Administration of the People 's Republic of China on October 24, 2014 approved its listing, the drug registration approval number: 2014S00506. According to the State Food and Drug Administration drug clinical approval requirements of this product need to carry out IV clinical research, the purpose is to examine the efficacy of drugs in a wide range of conditions and adverse reactions to evaluate the general or special population in the use of the interests and risks , To further observe the safety and efficacy of drugs.

ELIGIBILITY:
Inclusion Criteria:

* In line with the diagnosis of uterine fibroids;
* With fibroids associated with clinical symptoms (such as uterine bleeding symptoms, symptoms of oppression, pain symptoms, etc.); or nearly 3 months fibroids gradually grow; or the largest fibroid diameter ≥ 5cm;
* Women of childbearing age over 18 years of age;
* Voluntarily tested and signed informed consent

Exclusion Criteria:

* Unexplained or vaginal bleeding other than uterine fibroids;
* Combined with malignant tumors (including reproductive and other systems), or endometrial ≥ 17mm;
* Is the use of simple progesterone contraceptives, progesterone-containing intrauterine device or compound oral contraceptives;
* Is using ketoconazole, itraconazole, erythromycin, rifampicin, adrenocorticotropic hormone (hydrocortisone, prednisone, dexamethasone, etc.), and some anticonvulsants (phenytoin, Phenobarbital, carbamazepine), griseofulvin, nonsteroidal antiinflammatory drugs (aspirin, acetaminophen, ibuprofen, etc.) and can not be discontinued during the study;
* Pregnant women and lactating women and medication or medication within 3 months after the cessation of births;
* Severe heart, liver, kidney disease and adrenal insufficiency, and / or ALT, AST> 1.5 times the upper limit of normal, Cr> normal upper limit;
* Allergies or previous allergy to a variety of drugs, or the study of active ingredients in the medication or any excipient allergy;
* Patients who have participated in other clinical trials within 3 months;
* Other investigators who are not considered to be involved in this study.

Min Age: 18 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 434 (Actual)
Dates: Start 2017-06-01 (Actual); Primary Completion 2019-01-04 (Actual); Study Completion 2019-07-12 (Actual)

PRIMARY OUTCOMES:
Security assessments | Up to study completion at approximately 24 weeks
  Security assessments will include monitoring and recording all adverse events (AEs) and serious adverse events (SAEs).
Changes of uterine fibroids(maximal fibroids) | Through study completion，an average of half year
  Comparison of changes in the volume group of uterine fibroids (maximal fibroids)before and after treatment

SECONDARY OUTCOMES:
Comparison of changes in the uterine volume | Through study completion，an average of half year
  Comparison of changes in the uterine volume before and after treatment.
Comparison of the relevant indicators of anemia | Through study completion，an average of half year
  Before and after treatment on the relevant indicators of anemia(red blood cell count, erythrocyte ratio, hemoglobin) groups of visits to the relative baseline changes in the value of the description, the group comparison.
Evaluation of the uterine bleeding symptoms | Through study completion，an average of three months
  The uterine bleeding symptoms were recorded before treatment.
Operation situation(Perioperative transfusion improvement,Type of surgery) | Through study completion，an average of half year
  When surgery was occurred, recording perioperative blood transfusion values; if the operation was performed, the proportion of subjects using minimally invasive surgery was calculated for all subjects.
Clinical symptom scores | Through study completion，an average of half year
  The clinical symptom scores were recorded before treatment.

CONTACTS AND LOCATIONS:
Overall Officials: Yingfang Zhou, M.D., Principal Investigator — Beijing Univesitay First Hospital
Locations (26):
- China (26):
  - Beijing Maternal and Child Health Care Hospiatl of Capital Medical Hospital, Beijing, Beijing Municipality
  - Beijing University First Hospital, Beijing, Beijing Municipality
  - Fuling Center Hospital of Chongqing City, Chongqing, Chongqing Municipality
  - The Second Hospital of Chongqing Medical Universit, Chongqing, Chongqing Municipality
  - The Second Hospital of Logyan, Longyan, Fujian
  - Quanzhou First Hospital, Quanzhou, Fujian
  - Guangdong Hospital for Maternal amd Child Health Care, Guangdong, Guandong
  - The Third Affillated Hospital of Southern Medical University, Guangzhou, Guangdong
  - The Fouth Hospital of Shijiazhuang, Shijiazhuang, Hebei
  - The Second Affiliated Hospital of Harbin Medical Universty, Harbin, Heilongjiang
  - Huaihe Hospital of Henan University, Kaifeng, Henan
  - The Second Affillated Hoapital of Zhenghzou University, Zhengzhou, Henan
  - Tongji Hospital of Tongji Medical College of Huazhong Universty of Science and Technology, Wuhan, Hubei
  - Changsha Hospital for Maternal amd Child Health Care, Changsha, Hunan
  - Jiangxi Maternal and Child Health Hospital, Nanchang, Jiangxi
  - Weifang People's Hospital, Weifang, Shandong
  - Obstetrics and Gynecology Hospital of Fudan Universty, Shanghai, Shanghai Municipality
  - Shanghai TCM-INTEGATED Hospital,Shanghai University of TCM, Shanghai, Shanghai Municipality
  - Westnorth Matertal and Child Hospital, Xian, Shanxi
  - Yanan University Affillated Hospital, Yanan, Shanxi
  - Chendu Third Hospital, Chengdu, Sichuan
  - Chengdu Women and Chirdren's Central Hosptal, Chengdu, Sichuan
  - Mianyan Central Hospital, Mianyang, Sichuan
  - The First People's Hospital of Yibin, Yibin, Sichuan
  - Tianjin Central Hoapital of Gynecology Obstetrics, Tianjin, Tianjin Municipality
  - Women's Hospital of Zhejiang Medical University, Hangzhou, Zhejiang

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Shen Q, Hua Y, Jiang W, Zhang W, Chen M, Zhu X. Effects of mifepristone on uterine leiomyoma in premenopausal women: a meta-analysis. Fertil Steril. 2013 Dec;100(6):1722-6.e1-10. doi: 10.1016/j.fertnstert.2013.08.039. Epub 2013 Oct 2. PMID 24094421
- [Background] Wang H, Jin J. [Effects of mifepristone on estrogen and progestin receptors in human uterine leiomyoma]. Zhonghua Fu Chan Ke Za Zhi. 2000 Feb;35(2):79-81. Chinese. PMID 11809103
- [Background] Yang Y, Zheng S, Li K. [Treatment of uterine leiomyoma by two different doses of mifepristone]. Zhonghua Fu Chan Ke Za Zhi. 1996 Oct;31(10):624-6. Chinese. PMID 9275461
- [Background] Eisinger SH, Meldrum S, Fiscella K, le Roux HD, Guzick DS. Low-dose mifepristone for uterine leiomyomata. Obstet Gynecol. 2003 Feb;101(2):243-50. doi: 10.1016/s0029-7844(02)02511-5. PMID 12576246
- [Background] Eisinger SH, Bonfiglio T, Fiscella K, Meldrum S, Guzick DS. Twelve-month safety and efficacy of low-dose mifepristone for uterine myomas. J Minim Invasive Gynecol. 2005 May-Jun;12(3):227-33. doi: 10.1016/j.jmig.2005.01.022. PMID 15922980
- [Background] Kulshrestha V, Kriplani A, Agarwal N, Sareen N, Garg P, Hari S, Thulkar J. Low dose mifepristone in medical management of uterine leiomyoma - an experience from a tertiary care hospital from north India. Indian J Med Res. 2013 Jun;137(6):1154-62. PMID 23852296